CLINICAL TRIAL: NCT03666819
Title: Phase II Trial of CO2RE Laser for Patients With Stage 0-III Hormone Receptor-Positive Breast Cancer on Aromatase Inhibitors With Vulvovaginal Atrophy
Brief Title: Carbon Dioxide Fractional Laser in Treating Participants With Stage 0-III Hormone Receptor-Positive Breast Cancer With Vulvovaginal Atrophy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer will not be supporting this study
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1892; NCI-2018-01774 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1892 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2018-10

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Breast Adenocarcinoma; Dyspareunia; Estrogen Receptor Positive; Progesterone Receptor Positive; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Vaginal Dryness; Vaginal Itching; Vulvovaginal Atrophy
MeSH Terms: conditions — Breast Carcinoma In Situ; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (carbon dioxide fractional laser) (Experimental): Participants undergo carbon dioxide fractional laser therapy over 10-15 minutes on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: Carbon Dioxide Fractional Laser; Other: Questionnaire Administration

INTERVENTIONS:
Device: Carbon Dioxide Fractional Laser — Undergo CO2RE laser therapy
  Other Names: CO2 Fractional Laser
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well carbon dioxide fractional (CO2RE) laser works in treating participants with stage 0-III hormone receptor-positive breast cancer with vulvovaginal atrophy associated with dryness, inflammation or thinning of the epithelial lining of the vulva and vagina. CO2RE laser is a device that delivers controlled CO2 energy to the vaginal tissue and may help treat vaginal symptoms such as itching, burning, painful sexual intercourse, thickened or thin skin of the vulva, and stinging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the reduction in Vulvovaginal Symptom Questionnaire (VSQ) score at 3-month follow up after CO2RE laser treatment.

SECONDARY OBJECTIVES:

I. To evaluate the reduction in VSQ score after CO2RE laser treatment 6-month follow-up and 12-month follow-up.

II. To evaluate Female Sexual Function Index (FSFI) score before and after treatment with CO2RE laser.

III. To evaluate Urogenital Distress Inventory (UDI) 6 score before and after treatment with CO2RE laser.

IV. To evaluate vaginal health index score and vaginal caliber before and after treatment with CO2RE laser.

V. To evaluate discomfort and pain during CO2RE laser treatment using the visual analog scale.

VI. To evaluate treatment satisfaction after CO2RE laser treatment using 5-point Likert scale.

VII. To evaluate adherence to aromatase inhibitor at 6 and 12 months after CO2RE laser treatment.

EXPLORATORY OBJECTIVES:

I. To assess the change in the vaginal cytology using vaginal maturation index at baseline and during follow-up.

II. To assess serum estradiol level at baseline and after CO2RE laser treatment.

OUTLINE:

Participants undergo carbon dioxide fractional laser therapy over 10-15 minutes on day 1. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adenocarcinoma of the breast stage 0-III
* Evidence of hormone sensitivity with estrogen receptor (ER) and/or progesterone receptor (PR) positive >= 1% of primary tumor tissue
* Currently or will be starting on aromatase inhibitor (letrozole, anastrozole, or exemestane)
* Willingness to self-report vaginal itching, dryness, or dyspareunia
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Obtained =< 28 days prior to registration: Hemoglobin >= 8.0 g/dL
* Obtained =< 28 days prior to registration: Absolute neutrophil count (ANC) >= 1500/mm^3
* Obtained =< 28 days prior to registration: Platelet count >= 75,000/mm^3
* Obtained =< 28 days prior to registration: Total bilirubin =< 3.0 x upper limit of normal (ULN)
* Obtained =< 28 days prior to registration: Aspartate transaminase (AST) =< 3 x ULN
* Obtained =< 28 days prior to registration: Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 2 x ULN OR if patient is receiving anticoagulant therapy and PT/INR or partial thromboplastin time (PTT) is within therapeutic range of intended use of coagulants
* Obtained =< 28 days prior to registration: Calculated creatinine clearance =< 3 x ULN
* Recent negative Papanicolaou (PAP) smear within 1 year. In patients who do not have recent PAP smear, PAP smear should be obtained as per standard of care during the screening process prior to enrollment
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Previous use of CO2 fractional within 1 year
* Receiving any form of hormone replacement therapy, including topical estrogens, testosterone, and dehydroepiandrosterone (DHEA) or selective estrogen receptor modulator (SERM), including tamoxifen and ospemifene
* History of or current dysplastic nevi in the area that will be treated
* Prolapse uterus > stage II according to the International Continence Society pelvic organ prolapse quantification (ICS-POP-Q) system
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of the treatment
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy. NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Evidence of urinary tract infection (UTI) based on the urinalysis (UA) at the time of the screening. Patients with evidence of UTI can be enrolled after UTI is treated and repeated UA and/or urine culture shows no further evidence of ongoing infection
* Evidence of injuries, bleeding, or evidence suggestive of dysplasia in the external vaginal area or vaginal canal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in Vulvovaginal Symptom Questionnaire (VSQ) (symptoms, emotions, and life-impact) | Baseline up to 3 months
  Descriptive statistics (mean, standard deviation [SD], median, interquartile range [IQR]) using frequency table and histogram will be used to summarize the reduction in the sum of VSQ total score first three scales of the VSQ (symptoms, emotions, and life-impact) at 3 months after treatment versus (vs.) baseline.

SECONDARY OUTCOMES:
Reduction in VSQ score (symptoms, emotions, and life-impact) | Baseline up to 12 months
  Will evaluate the sum of first three scales of the VSQ (symptoms, emotions, and life impact), VSQ total scale, and sub-scales. Descriptive statistics (mean, SD, median, IQR) and longitudinal plots (raw value, change, change in percentage) will be used to summarize the sum of VSQ total score first three scales of the VSQ (symptoms, emotions, and life-impact), VSQ total scale and subscales.
Female Sexual Function Index (FSFI) score | Baseline up to 12 months
  Descriptive statistics (mean, SD, median, IQR) and will be used to summarize FSFI total score and subscales before and after treatment.
Urogenital Distress Inventory (UDI) 6 score | Baseline up to 12 months
  Descriptive statistics (mean, SD, median, IQR) and will be used to summarize UDI-6 score before and after treatment.
Vaginal health index score | Baseline up to 12 months
  Descriptive statistics (frequency table) and histogram will be used to summarize vaginal health index score before and after treatment.
Vaginal caliber | Baseline up to 12 months
  Descriptive statistics (mean, SD, median, IQR) and will be used to summarize vaginal caliber before and after treatment.
Discomfort and pain during carbon dioxide fractional (CO2RE) laser treatment using the visual analog scale | Up to 12 months
  Descriptive statistics (mean, SD, median, IQR) and will be used to summarize the visual analogue pain scale during treatment.
Treatment satisfaction as measured by 5-point Likert scale | Up to 12 months
  Descriptive statistics (frequency table) and histogram will be used to summarize treatment satisfaction after CO2RE laser treatment using 5-point Likert scale during follow-up
Adherence to aromatase inhibitor as measured by the Simplified Medication Adherence Questionnaire | Up to 12 months
  Descriptive statistics (frequency table) and histogram will be used to summarize the Simplified Medication Adherence Questionnaire during follow-up.
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 12 months
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns.

OTHER OUTCOMES:
Change in vaginal cytology using vaginal maturation index | Baseline up to 12 months
  Descriptive statistics (mean, SD, median, IQR) and longitudinal plots (raw value, change, change in percentage) will be used to summarize the change in the vaginal cytology using vaginal maturation index.
Assessment of serum estradiol levels | Baseline up to 12 months
  Descriptive statistics (mean, SD, median, IQR) and longitudinal plots (raw value, change, change in percentage) will be used to summarize serum estradiol level at baseline and after CO2RE laser treatment and the change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, Principal Investigator — Mayo Clinic